CLINICAL TRIAL: NCT01623960
Title: A Nationwide Multicenter Study on the Quality of Life in Adult Patients With Severe Haemophilia in Turkey
Brief Title: Quality of Life in Adult Patients With Severe Haemophilia in Turkey
Acronym: TurkHaemQoL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Turkish Society of Hematology (Other)
Responsible Party: Principal Investigator, M. Cem Ar, Member, Subcommittee of Haemophilia, Turkish Society of Haematology, Turkish Society of Hematology
Other Study IDs: THD-HAEM-QoL
Record Dates: First submitted 2012-06-17; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Haemophilia
Keywords: severe haemophilia; quality of life
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary aim of this study is to evaluate the overall quality of life in adult patients with severe haemophilia (an inherited bleeding disorder affecting mainly men) in Turkey and to assess the impact of certain disease and drug related factors (treatment modality, presence of viral disease, inhibitor, etc.) on the quality of life.

DETAILED DESCRIPTION:
Haemophilia is an inherited bleeding disorder affecting one in 10000 male births worldwide. People with severe haemophilia usually suffer from recurrent life threatening bleeds (e.g. into the brain, digestive system or abdomen) and/or disabling degenerative disease of weight bearing joints (e.g. knees, elbows and ankles)resulting from haemorrhage into the joints. Daily activities of people with haemophilia has been shown to be dramatically hampered by the resultant joint damage. Evaluation of quality of life issues in people with severe haemophilia would help to create awareness of their problems and limitations. This would also set up the scene for developing policies to improve the treatment options/facilities and social life of the patients. Current study aims to assess the quality of life of adult patients with severe haemophilia in a developing country (Turkey) by using a validated Quality of Life Questionnaire (Turkish version of Haem-A-QoL).

ELIGIBILITY:
Inclusion Criteria:

* age equal or greater than 18 years
* male gender
* factor VIII or IX level equal or below 1%
* patients that are willing to participate and have given a written consent

Exclusion Criteria:

* age less than 18 years
* females
* factor levels above 1%

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male patient with severe haemophilia followed at 10 different haemophilia centers in Turkey
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-02 (Estimated)